CLINICAL TRIAL: NCT03404102
Title: Discontinuation Rates Among Copper Intrauterine Device Users in Primary Healthcare Unit and University Clinic. Is There a Difference?
Brief Title: Discontinuation Rate Among Copper IUD Users
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: noha mohamed elzaydy (Other)
Responsible Party: Sponsor-Investigator, noha mohamed elzaydy, researcher, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: Cu-IUD
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Contraceptive Device; Intrauterine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- university clinic: * Enrollment: 200 Subjects will be enrolled from women attending family planning clinic for Cu- IUD insertion
  * Informed Consent: All participants will give their informed consent prior to enrollment.
  * Data collection & recording: Data of each patient will be recorded in a Case Record Form (CRF).
  * Follow up visits /questionnaire: will be conducted from each subject at 6 months and 12 months after Cu-IUD insertion. User satisfaction score and haemoglobin serum level will be included in the questionnaire.
  Interventions: Device: Cu-IUD
- primary healthcare unit clinic: * Enrollment: 200 Subjects will be enrolled from women attending family planning clinic for Cu- IUD insertion
  * Informed Consent: All participants will give their informed consent prior to enrollment.
  * Data collection & recording: Data of each patient will be recorded in a Case Record Form (CRF).
  * Follow up visits /questionnaire: will be conducted from each subject at 6 months and 12 months after Cu-IUD insertion. User satisfaction score and haemoglobin serum level will be included in the questionnaire.
  Interventions: Device: Cu-IUD

INTERVENTIONS:
Device: Cu-IUD — Copper Intra-uterine device used as contraceptive method

SUMMARY:
The intrauterine device (IUD) is one of the most widely used reversible, long-term contraceptive methods in the world. But despite all its advantages; discontinuation rate of IUD ranged from 9.6% to 37.3 % (according to Demographic and Health Surveys data). In Egypt, in 2014, the discontinuation rate of IUD (within 12 months of use) was 14.3%.This study explores the differences around this rate in Egyptian university clinic and primary healthcare clinic with detailed percentages of possible causes.

DETAILED DESCRIPTION:
The aim of the study is to compare between primary health care unit and university family planning clinic in discontinuation rate among copper IUD users.

1. The Research Hypothesis: (Null hypothesis)

   • In women using copper IUD, discontinuation rate in primary health care unit and university clinic may be similar.
2. The Research Question:

   • In women using copper IUD, Does discontinuation rate in primary health care unit and university clinic differ?
3. METHODOLOGY:

Patients and Methods

• Study setting:

* Family planning Outpatient clinic of Ain Shams Maternity Hospital, (ASUMH)
* primary health care unit in ain shams area

  • Study population:
* Study period: 1 year
* Sample size: was calculated using Sample size computer program 11. After review of literature, no previous similar study was done before, so assume a discontinuation rate of 50% among Cu-IUD users in primary healthcare unit and 25% among Cu-IUD users in university clinic. Based on these values; the study will include 170 Cu-IUD users; equally selected as 85 subjects from each clinic. But due to the expected drop outs, recruitment will start by 200 women from each clinic.

  * Statistics:

    * Descriptive statistics for measured variables will be expressed as range, mean and standard deviation (for metric data); range, median and interquartile range (for discrete data); and number and proportions (for categorical data). Cu-IUD discontinuation findings in each clinic will be compared using the t-test or the Mann-whitney U test depending on whether the measured parameters are guassian variables. A P-value of 0.05 or less will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age from 18-49 years. 2. Women planning for Cu-IUD insertion as a contraceptive method.

Exclusion Criteria:

* 1. Any woman with condition included in Category 3 or 4 for Cu-IUD in medical eligibility criteria for contraceptive use (MEC) -World Health Organization-2015.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women attending family planning for Cu- IUD insertion who meet inclusion criteria
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
measure discontinuation rate | 1 year
  • To measure the discontinuation rate among copper IUD users in primary health care unit and university clinic.

SECONDARY OUTCOMES:
exclude anemia | 1 year
  To exclude Anemia from reasons of Cu-IUD discontinuation.
comparison | 1 year
  • To identify reasons of discontinuation among Copper IUD users and percentage of each cause in both university clinic and primary health care unit.
users" satisfaction | 1 year
  • To measure copper IUD users' satisfaction of this contraceptive method in both university clinic and primary health care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Ain Shams Maternity Hospital, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity hospital, Cairo, Ain Shams, Egypt

IPD SHARING:
Plan to Share IPD: Undecided